CLINICAL TRIAL: NCT02677129
Title: Physical Function and Activities of Daily Living in Cancer Patients During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Agaplesion Markus Krankenhaus gGmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPM2015-003
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Advanced Gastrointestinal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- home-based exercise intervention (Experimental): home-based exercise intervention:
  Endurance training (moderate intensity; walking), 3-5 times per week Patients will receive exercise counselling how to realize the planned intervention home-based. Further, they will be asked to fill out an exercise log. The study team will periodically review adherence to the intervention and identify problems.
  Interventions: Other: home-based exercise intervention
- Waiting control group (No Intervention): The wait list control group receives usual care over the study period. Usual care depends on the hospital guidelines as well as oncologists' and physicians' consideration.

INTERVENTIONS:
Other: home-based exercise intervention — Endurance training (moderate intensity; walking), 3-5 times per week Patients will receive exercise counselling how to realize the planned intervention home-based. Further, they will be asked to fill out an exercise log. The study team will periodically review adherence to the intervention and identify problems.
  Arms: home-based exercise intervention

SUMMARY:
The study is a randomized controlled trial with the aim to examine the feasibility and the effects of a home-based exercise intervention program on activities of daily living (ADL) in patients with advanced gastrointestinal cancer undergoing chemotherapeutic treatment. Further outcomes include functional and body status, quality of life, body composition, and chemotherapy completion rate. Study participants will be randomized to an exercise intervention group or a wait-list control group

DETAILED DESCRIPTION:
A randomised longitudinal study. A total of 44 gastrointestinal cancer patients before their first-line chemotherapy are recruited and randomised into one of two treatment groups A: Home based- physical activity or B: wait-control. The intervention period is 12 weeks. Primary outcome are the ADLs (iADL 1-8; FIM 1-7).Secondary outcomes are the physical activity, quality of life, peripheral polyneuropathy, chemotherapy regimen, gait speed, postural stability, maximal isometric voluntary force of the upper extremity, Maximal isometric voluntary force (MIVF) and strength endurance of the lower extremity, nutritional state, body composition and perceive functional ability. All measurements are standardized and are performed before chemotherapy, after 2 cycles of chemotherapy (4-6weeks) and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically classified gastrointestinal cancer
* UICC III-IV
* Prior to (planned) first-line chemotherapy (curative und palliative)
* ≥50 years

Exclusion Criteria:

* ECOG > 2
* Systemic diseases (MS, ALS)
* disorders (neurological, skeletal, muscular, mental or cognitive) or drug use (irrespective of the cancer therapy) that may affect gait, balance or muscular strength
* chronic infection, uncontrolled hypertension (diastolic pressure over 95 mmHg)
* vestibulopathies
* uncorrected visual deficits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Change between the first 12 weeks of chemotherapy
  Short battery of physical performance tests used to assess lower extremity function. Balance, gait, strength, and endurance are evaluated.

SECONDARY OUTCOMES:
Daily physical activity | 3 times in the course of 12 weeks of chemotherapy
  7 days accelerometry
Polyneuropathy | 3 times in the course of 12 weeks of chemotherapy
  Measuring the sensibility with a Rydel-Seiffer tuning fork
Gait speed | 3 times in the course of 12 weeks of chemotherapy
  usual gait speed (km/h) on a capacitive force-measuring platform (30Hz) WinFDM v0.0.41® (Zebris© GmbH, Isny, Germany)
Postural sway | 3 times in the course of 12 weeks of chemotherapy
  balance measuring (COP) on a capacitive force-measuring platform (30Hz) WinFDM v0.0.41® (Zebris© GmbH, Isny, Germany)
Maximum isometric voluntary force of the upper extremity | 3 times in the course of 12 weeks of chemotherapy
  JAMAR Hand Dynamometer
Maximum isometric voluntary force of the lower extremity | 3 times in the course of 12 weeks of chemotherapy
  The maximal isometric voluntary force (MIVF) of the randomly chosen knee extensor is measured with a strain gauge force transducer (ASYS®; SPOREG; 100 Hz) in a standardised seating position (predefined knee and hip angle = 90°).
Muscular endurance (Chair-Rise Test) | 3 times in the course of 12 weeks of chemotherapy
  For the five times sit to stand test patients start in a standard position sitting on a chair that is placed next to the wall with the arms folded across their chest. They are asked to stand up from a chair to a full standing position and sit down again keeping the arms crossed for five times as quickly as possible.
Quality of life | 3 times in the course of 12 weeks of chemotherapy
  European Organisation for Research and Treatment of Cancer (EORTC_QLQ-C30)
Quality of life | 3 times in the course of 12 weeks of chemotherapy
  The 36-Items Short Form Health Survey (SF-36)
Nutrition Assessment | 3 times in the course of 12 weeks of chemotherapy
  Mini Nutritional Assessment (MNA)
Phase angle | 3 times in the course of 12 weeks of chemotherapy
  multifrequent bioelectrical impedance analysis (DATA-Input) measuring the phase angle
Body cell mass | 3 times in the course of 12 weeks of chemotherapy
  multifrequent bioelectrical impedance analysis (DATA-Input) measuring the body cell mass (BCM)
Fat mass | 3 times in the course of 12 weeks of chemotherapy
  multifrequent bioelectrical impedance analysis (DATA-Input) measuring the fat mass
Perceived functional ability | 3 times in the course of 12 weeks of chemotherapy
  perceived functional ability scale
Activities of daily living | Change between the first 12 weeks of chemotherapy
  Functional Independence Measurement (FIM) Questionnaire
Activities of daily living | Change between the first 12 weeks of chemotherapy
  - instrumental Activity of Daily Living (iADL)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Banzer, Prof., Principal Investigator — Department of Sports Medicine, Goethe University Frankfurt
Locations (1):
- Agaplesion Markus Hospital, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No
Only pseudonymised data without the plan to share